CLINICAL TRIAL: NCT03840070
Title: A Single-center, Open-label, Long-term, Exploratory Study to Determine the Efficacy and Safety of Repeat-dose Potenfill for Temporary Penile Enhancement
Brief Title: The Efficacy and Safety of Repeat-dose Potenfill for Temporary Penile Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT05-KR18PGE1005
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Penile Girth Enhancement; Penile Enhancement

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Potenfill (Experimental)
  Interventions: Device: Potenfill

INTERVENTIONS:
Device: Potenfill — Maximum: 22ml
  Other Names: hyaluronic acid filler

SUMMARY:
This clinical study is for small-penis syndrome males who have previously been treated with hyaluronic acid filler for the purpose of increasing their penis.

This study will determine the long-term efficacy and safety of Potenfill.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged above 19 and below 65. (20≤male≥65)
* Subjects will sign an informed consent form

Exclusion Criteria:

* Prior treatment for penile enhancement (e.g. fat, dermal graft).
* Allergic to hyalluronic acid.

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Subject satisfaction on the penile appearance at 12 months after application of Potenfill | 12 month
  Satisfaction with the physical appearance of penis as assessed by the subject at 12 months after the application of investigational medical device.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea university guro hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided